CLINICAL TRIAL: NCT05418140
Title: Adenomyosis and Pregnancy Outcomes in Women Undergoing Assisted Reproductive Technology Treatment: a Prospective Multicentre Cohort Study (AdAPT-ART)
Brief Title: Adenomyosis and Pregnancy Outcomes in Women Undergoing Assisted Reproductive Technology Treatment
Acronym: AdAPT-ART
Status: Active, not recruiting | Type: Observational
Sponsor: CARE Fertility UK (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: AdAPT-ART
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-04

CONDITIONS: Adenomyosis; Infertility; ART; Pregnancy Loss; Miscarriage
Keywords: Adenomyosis; Infertility; ART
MeSH Terms: conditions — Adenomyosis; Infertility; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women with diagnosis of adenomyosis on ultrasound scan: The cohort group (375 participants) will comprise of women diagnosed with adenomyosis on pre-treatment baseline ultrasound scan before ART treatment who satisfy the eligibility criteria and consent to participate in the study.
  September 2022: Amendments to the protocol: Some of the methodological aspects of the AdAPT-ART study have been revisited to ensure timely delivery of the study to a full sample size. These amendments have been approved by the local ethics committee.
  Amendment sample size:
  Sample size of 276 women with adenomyosis and 552 women with normal uterus with 2:1 control: cohort design. Power remains 80%
  Interventions: Other: Ultrasound diagnosis of adenomyosis
- Control group: Women with normal uterus on baseline ultrasound scan: Women with normal uterus on baseline ultrasound scan during the study duration will be used as control (375 participants) and will be matched for the following variables: age, embryo quality, type of ART cycle (donor or self and IVF or ICSI) and number of embryos transferred. The eligibility criteria will be applicable to the controls as well.
  September 2022: Amendments to the protocol: Some of the methodological aspects of the AdAPT-ART study have been revisited to ensure timely delivery of the study to a full sample size. These amendments have been approved by the local ethics committee.
  Amendment sample size:
  Sample size of 276 women with adenomyosis and 552 women with normal uterus with 2:1 control: cohort design. Power remains 80%
  Interventions: Other: Ultrasound diagnosis of adenomyosis

INTERVENTIONS:
Other: Ultrasound diagnosis of adenomyosis — The diagnosis of adenomyosis will be made using transvaginal ultrasound scan (TVS) (2D and 3D Ultrasound and applying Morphological Uterus Sonographic Assessment (MUSA) criteria (Van den Bosch et al, 2015).

SUMMARY:
Rationale: A rising number of adenomyosis cases are being diagnosed in women in the age group of 30 to 40 years. This is due to a combination of better diagnostic imaging techniques and a higher number of women delaying the fulfilment of their fertility aspirations. The association between adenomyosis and pregnancy outcomes in women with subfertility has not been adequately explained by existing evidence due to lack of data on the association between the severity of adenomyosis, disease location, presence of symptoms and coexisting gynaecological conditions and pregnancy loss in women undergoing fertility treatment. There is a need to improve our understanding of prognostic features which would be beneficial in counselling women with adenomyosis undergoing fertility treatment and inform future management options. The investigators propose a research body of work aimed at improving our understanding of adenomyosis and its association with pregnancy loss. Objective: The aim of the study is to determine the association between adenomyosis and pregnancy loss in women undergoing assisted reproductive technology (ART) treatment. Study design: Prospective multicentre cohort study. The cohort will comprise of women with adenomyosis undergoing ART treatment and the control group will include women with normal uterus on baseline ultrasound scan undergoing ART treatment during the study duration. Settings: The study will be conducted at all main CARE fertility units, one of the largest providers of fertility treatment in the United Kingdom. Participant population with exposure and sample size: The cohort group will comprise of women diagnosed with adenomyosis on pre-treatment baseline ultrasound scan before ART treatment who satisfy the eligibility criteria and consent to participate in the study. The total sample size for this study will be 750 participants with 375 women in each arm. Recruitment will take place over the course of 18 months. Diagnostic tool for detection of exposure: The diagnosis of adenomyosis will be made using transvaginal ultrasound scan (TVS) (2D and 3D Ultrasound and applying Morphological Uterus Sonographic Assessment (MUSA) criteria. Schematic mapping system of adenomyosis severity proposed by Lazzeri and colleagues will be used to grade the severity of adenomyosis. Eligibility: Inclusion criteria: All women aged >18 years and ≤42 years undergoing IVF/ICSI cycle. Exclusion criteria: Women with coexisting fibroid uterus, endometrioma confirmed on USS or known laparoscopic diagnosis of endometriosis (with histological confirmation), untreated hydrosalpinx, uterine malformation, previous myomectomy, previous surgery for adenomyosis or inconclusive USS. Recruitment: All women undergoing pre-treatment pelvic ultrasound scans before ART treatment will be screened for adenomyosis at the participating centres. Women who meet the eligibility criteria will be provided with an information leaflet about the study. They will be enrolled in the study after informed consent is obtained. The severity of adenomyosis will be subsequently evaluated using stored 2D and 3D ultrasound scan (USS) images. Several demographic, clinical and treatment characteristics will be recorded for each participant. Control: To ensure adequate comparability of the cohort, women with normal uterus on baseline ultrasound scan during the study duration will be used as control and will be matched for the following variables: age, embryo quality, type of ART cycle (donor or self and IVF or ICSI) and number of embryos transferred. The eligibility criteria will be applicable to the controls as well. Outcome measures: Primary outcome: Pregnancy loss up to 24 weeks out of all pregnancies achieved. The pregnancy loss will include biochemical pregnancy loss, miscarriage, pregnancy of unknown location (PUL) and ectopic pregnancy. This will be reported per embryo transfer and per woman. Secondary outcomes:1. Implantation rate per embryo transfer (number of gestational sacs divided by number of embryos transferred) and per woman; 2. Biochemical pregnancy rate per embryo transfer (positive pregnancy test following embryo transfer) and per woman; 3. Clinical pregnancy rate per embryo transfer (presence of at least one intrauterine gestational sac on ultrasound) and per woman; 4. Ongoing pregnancy rate per woman (defined as a live pregnancy at 12 weeks onwards); 5. Live birth rate after 34 weeks per woman. Subgroup analysis: We will carry out subgroup analysis according to specific patient characteristics. These analyses will include, but not necessarily be limited to women with the following characteristics:1. Varying severity of adenomyosis; 2. Presence /absence of symptoms of adenomyosis; 3. Frozen vs. Fresh embryo transfer; 4. Short vs. long vs. ultralong ovarian stimulation protocol; 5. Recurrent miscarriages; 6. Other associations that may become apparent in post-hoc analyses.

DETAILED DESCRIPTION:
The study investigators propose a prospective observational study to determine the association between adenomyosis and pregnancy loss in women undergoing ART treatment using a consistent classification system for adenomyosis diagnosed on ultrasound scan. This will be supplemented with subgroup analyses such as the following: presence vs absence of adenomyosis symptoms; frozen and fresh embryo transfer cycles; and varying severity of adenomyosis. These subgroup analyses will help determine the influence of these factors on the association between adenomyosis and pregnancy outcomes.

AIMS AND OBJECTIVES

AIM OF THE STUDY: To investigate the association between adenomyosis and pregnancy outcomes in women undergoing ART treatment.

PRIMARY OBJECTIVES: To compare the incidence of pregnancy loss in women with and without adenomyosis undergoing ART treatment. The pregnancy loss will include biochemical pregnancy loss, miscarriage, pregnancy of unknown location (PUL) and ectopic pregnancy.

SECONDARY OBJECTIVES:

* To compare rates of treatment outcomes (implantation rate, biochemical pregnancy rate, clinical pregnancy rate, ongoing pregnancy rate, and live birth rate) in women with and without adenomyosis undergoing ART treatment.
* To investigate whether there is an association between the severity of adenomyosis and pregnancy outcomes

STUDY DESIGN AND SETTING

STUDY DESIGN: Prospective multicentre cohort study SETTING The study will be conducted at all main CARE fertility units, one of the largest providers of fertility treatment, in the United Kingdom.

PARTICIPANT POPULATION

* Population: The study cohort will comprise of women diagnosed with adenomyosis on pre-treatment baseline ultrasound scan before ART treatment who satisfy the eligibility criteria and consent to participate in the study.
* Duration of recruitment: Recruitment will take place over the course of 18 months
* Sample size: The total number of participants required to determine the association between women with adenomyosis and the primary outcome (pregnancy loss) will be 750 with 375 participants per arm. This will ensure that the study is powered to 80%. The estimated sample size for a two-sample proportions was calculated using Stata 17.0. The basis for this calculation stems from a recent meta-analysis which showed a miscarriage rate of 31.33% among women with adenomyosis. To detect a 9.53% increase in miscarriage from the baseline risk of 21.8% in women undergoing ART treatment, 337 clinical pregnancies will be needed (alpha error: 0.05, beta error: 0.2, power 80%). Anticipating a 10% loss to follow up and inconclusive USS diagnosis, total number of participants per arm required will be 375 (374.44). This has been further elaborated in the statistics section of this study protocol.
* Control: To ensure adequate comparability of the cohort, women with a normal uterus on baseline ultrasound scan for the duration of the study will be used as controls and will be retrospectively matched for the following variables: age, embryo quality, type of ART cycle (donor or self and IVF or ICSI) and number of embryos transferred. The eligibility criteria will be applicable to the control group as well.
* Blinding: Women will be screened for adenomyosis during the pre-treatment baseline ultrasound scan (USS) and there will be no formal endeavour to blind the USS operators to the baseline characteristics of the women. All the stored ultrasound images of adenomyotic and normal uteruses will be reviewed by a 2nd clinician who will be blinded to the baseline characteristics of the women to avoid identification and recruitment bias. ART cycle management will be as per standard protocol with no blinding of the treating clinician to the diagnosis of adenomyosis. A pre-specified subgroup analysis for study population with different types of stimulation protocol will be performed. Since the primary outcome measurement will be USS based, there will not be any blinding of the outcome assessors.

DIAGNOSTIC TOOL FOR DETECTION OF EXPOSURE

* Diagnostic tool: The pooled sensitivity and specificity of TVUS for the diagnosis of adenomyosis for all combined imaging characteristics is 83.8% and 63.9% for 2D and 88.9% and 56.0% for 3D, respectively. The diagnosis of adenomyosis in the study participants will be made using transvaginal ultrasound scan; 2D and 3D Ultrasound with a 4-9 MHz trans-vaginal probe on Voluson S8.
* Pre-implementation meeting: Preliminary meetings to discuss the sonographic appearance and diagnostic criteria for adenomyosis will be organised with the clinicians and nurse sonographers participating in the study. An operations manual will be disseminated to the participating centres to assure a uniform and standardised approach is followed for the diagnosis of adenomyosis.
* Timing of the diagnosis: At the time of baseline pre-treatment scan
* Image: Images will be printed or stored as 2D and 3D images. Where possible 2D video clips and 3D volumes will be stored as well
* Reliability assessment: Intra-observer reliability will be assessed using test-retest measure
* Diagnostic criteria: The Morphological Uterus Sonographic Assessment (MUSA) criteria will be used to describe the ultrasound features of adenomyosis. The MUSA criteria outlines the ultrasound features of myometrium and myometrial lesions using standardised terms, definitions and measurements. The MUSA criteria for diagnosis of adenomyosis on ultrasound is based on consensus opinion of a panel of clinicians with expertise in gynaecological ultrasonography, fertility treatment, hysteroscopy, general gynaecology and clinical research. A diagnosis of adenomyosis is made if any morphological features of adenomyosis are present. This stems from data demonstrating a strong correlation between the presence of at least one sonographic feature of adenomyosis with histopathological findings of adenomyosis. All the images stored will be re-reviewed by a 2nd clinician specialising in gynaecological ultrasound. Where the two practitioners do not reach a consensus on the diagnosis of adenomyosis, arbitration will be undertaken by a senior third clinician. If there is no consensus reached, the case will be excluded. The following MUSA criteria would be used for diagnosis of adenomyosis

  * Anteroposterior asymmetrical myometrial wall: Ratio of two walls above/below 1 or subjective impression. The anterior and posterior myometrial walls are measured from the external uterine serosa to the external endometrial contour. This should include the junctional zone (JZ) but not the endometrium and be perpendicular to the endometrium
  * Myometrial echogenicity: Overall heterogenous myometrium with fan shaped shadowing
  * Myometrial or sub-endometrial lesions: Myometrial cysts or Hyperechogenic islands or sub-endometrial echogenic lines/buds or fan shaped shadowing due to lesions
  * Junctional Zone (JZ): Thickened or irregular or interrupted or ill-defined
  * Vascularity of myometrial lesion: Translesional vascularity. In adenomyoma and focal adenomyotic lesions diffuse minimal vascularity seen as diffuse spread of small vessels within the myometrium. Translesional vascularity: defined as vessels perpendicular to the endometrium crossing the lesion.
  * Uterine contour: Globally enlarged uterus. Fundus of the uterus appears enlarged
* Classification of severity: A schematic mapping system of adenomyosis severity will be used for determining the severity of uterine adenomyosis. This has been chosen due to reproducibility, substantial to almost perfect interobserver agreement rate and clinical correlation with symptom severity. A score ranging from to 1 to 4 is attributed to each grade, and the sum of the score numbers is used to calculate the extension of the disease: mild (range, 1-3), moderate (4-6), and severe (>7). The investigators will also classify the extent of affected myometrial as a percentage: Mild (<25%), Moderate (25-50%), Severe (>50%). Stored 2D and 3D USS images of patients diagnosed with adenomyosis on USS will be reviewed by two clinicians to determine the severity score.

CONSENT Written informed voluntary consent will be obtained by the investigator for each potential participant meeting the diagnostic and eligibility criteria. Responsibility for taking consent will be either of a clinician or nurse as delegated by the Principal Investigator. To facilitate the consent process, each participant will be provided with a Participant Information Sheet (PIS). Adequate explanation about the purpose of the study, the exposure and possible benefits of the study will be discussed with each participant. The voluntary nature of the participation will be discussed. Participants will be informed that they may decline participation or withdraw from the study at any time without giving any reason. This will not affect their medical care or legal rights. Time will be given to the participants to read the PIS and to discuss their participation with others outside of the site research team. The participants will have the opportunity to ask questions before signing the latest version of the Informed Consent Form (ICF).

After the participant has signed and dated the consent form, the investigator or delegate will also sign and date the ICF. The consent signing will be done online where possible. There will be triplicates of the ICF; one copy will be given to the participant; a second copy will be filed in the woman's medical notes; and the original will be placed in the Investigator Site File (ISF). The participant will have the opportunity to ask questions about the study throughout the study duration. The record of the details of informed consent discussions will be made in the participant's medical notes. This will include the name of the study, date of discussion, summary of discussion, version number of the PIS given to participant and version number of ICF signed and date consent received.

RECRUITMENT AND ENROLMENT

All women undergoing pelvic pre-treatment ultrasound scans before fertility treatment will be screened for adenomyosis at the participating centres by the clinicians and nurses experienced in performing ultrasound scan. The clinicians and nurses will be performing the baseline scan as per the standard protocol and therefore blinding to the baseline characteristics of the women will not be possible. All the stored ultrasound images of adenomyotic and normal uterus will be reviewed by a 2nd clinician who will be blinded to the baseline characteristics of the women to avoid identification and recruitment bias. Women who meet the eligibility criteria will be provided with a PIS describing the study. They will be enrolled in the study after informed consent is obtained. The demographic, clinical and treatment characteristics which will be recorded and used for data analysis are outlined as below:

* Demographics: Age (in years), Ethnicity, BMI (in Kg/m2), Duration of subfertility, Ovarian reserve (AMH and AFC), Smoking/Alcohol intake
* Clinical history: Cause of subfertility, Associated male subfertility, Primary/Secondary subfertility, Presence/absence of symptoms of abnormal uterine bleeding, gynaecological pain symptoms, dysuria, dyschezia, Previous obstetric history (live birth, miscarriage).
* ART: IVF, ICSI, Previous number of IVF/ICSI cycles
* IVF cycle details: Type of ovarian stimulation protocol, Total Gonadotrophin dose and duration of stimulation, Number of mature follicles >14mm, Number of oocytes retrieved Metaphase 2 oocytes, Embryo quality, Fresh/Frozen embryo transfer, Endometrial preparation, Number of Embryos transferred, Day of embryo transfer, Thickness of endometrium

MANAGEMENT OF IVF/ICSI CYCLE FOR PARTICIPANT POPULATION Women recruited for the study will be offered ART treatment according to a standardised clinical protocol at CARE fertility. The starting dose of gonadotrophins and the type of protocol for stimulation will be based on patient's age, body mass index (BMI), AMH and the number of basal antral follicles. Transvaginal ultrasound and oestradiol measurements will be used to monitor follicular growth, and the doses of gonadotrophin will be adjusted accordingly. Trigger in form of HCG/ GnRH agonist will be given once at least two follicles are observed to be greater than 17 mm in diameter on ultrasound examination and oocyte retrieval will be carried out 36 h after injection of trigger. Embryo transfer will be carried out on day 2, day 3 or day 5 depending on the number of good quality embryo and the number of embryos transferred will be 1 or 2 depending on the age of the patient and the quality of embryo.

Since this study also includes frozen embryo transfer cycles, endometrial preparation will be as per FET protocols according to local practice (natural, stimulated, modified natural with HCG trigger, or hormone replacement therapy [HRT] cycles). All embryo transfers will be performed under transabdominal USS guidance using soft Wallace catheter. This will be followed by luteal phase support with progesterone (vaginal capsules at a dose of 400 mg twice daily or combined vaginal and subcutaneous progesterone at a dose of 25 mg once daily) until 8-12 completed weeks of gestation.

OUTCOME All women will be followed up for primary and secondary outcomes. The CARE Fertility electronic patient database will be used to record the outcome data and collated for subsequent analyses.

DATA HANDLING AND RECORD KEEPING Data will be stored in the CARE Fertility electronic patient record system in accordance with the Data Protection Act 2018. Patient data will be anonymised for the purposes of statistical analysis.

QUALITY CONTROL AND QUALITY ASSURANCE Principles of Good Clinical Practice will be followed throughout the study duration.

ADVERSE EVENT REPORTING Considering the observational nature of the study and no additional step involved in the study design other than baseline USS, there are no safety considerations involved.

STATISTICS

* SAMPLE SIZE The total number of participants required to determine the association between adenomyosis and the primary outcome (miscarriage) would be 750 with 375 participant population per arm. This would ensure our study is powered to 80%. The estimated sample size for a two-sample proportions using two-sided test is calculated using Stata 17.0. The following explanation outlines the basis for the calculation: A recent meta-analysis has shown that the miscarriage rate among women with adenomyosis was 31.33%. The baseline risk of miscarriage in women undergoing ART treatment is 21.8%. To detect a 9.53% difference in incidence of miscarriage, 337 clinical pregnancies will be required per arm (alpha error: 0.05, beta error: 0.2, power 80%). Anticipating a 10% loss to follow up and inconclusive USS diagnosis, total number of participants per arm required will be 375 (374.44).
* OUTCOME MEASURE ANALYSIS The demographic, clinical and ART cycle characteristic comparison between group with adenomyosis and the control group will be completed using descriptive statistics. Categorical variables will be reported as frequencies and percentage and continuous variables as mean and standard deviation for normally distributed data. The Shapiro Wilk test will be used to determine the distribution of the data. Univariate analysis will be performed by using the student's t-test or Wilcoxon test for continuous variables and Chi square test or Fisher's exact test for categorical variables where appropriate.

The cohort group will comprise of women with USS diagnosis of adenomyosis and the control group will comprise of women with normal uterus on USS. The cohort and the control group will be matched for the following variables: age, embryo quality, type of ART cycle (donor or self and IVF or ICSI) and number of embryos transferred. Pregnancy outcomes will be reported as dichotomous variables. Generalised linear models will be used to determine the strength of the association between adenomyosis and pregnancy outcomes and will be reported as point estimates (e.g. risk ratios, odds ratios, risk differences) with 95% confidence interval. Generalised linear models with a binomial distribution with appropriate link functions will be used to calculate the adjusted relative risk and the mean differences, accounting for the following variables: BMI, ovarian reserve, previous IVF cycles, stimulation protocol, endometrial preparation and endometrial thickness prior to transfer. Statistical confidence will be determined by using the p value. Statistical analysis will be conducted using Stata 17.0.

• SUBGROUP ANALYSIS

A subgroup analysis for the primary outcome will also be conducted for women with:

* varying severity of adenomyosis
* presence /absence of symptoms of adenomyosis
* frozen vs fresh embryo transfer
* short vs. long vs. ultralong ovarian stimulation protocol
* recurrent miscarriages: loss of two or more pregnancies prior to 24 weeks of gestation as defined in the ESHRE guideline on recurrent pregnancy loss, 2018.
* other associations that may become apparent in post-hoc analyses. The subgroup characteristics will be described in detail and statistical analysis that has been outlined for the primary outcome will be followed for subgroup analysis

  * MISSING DATA AND ANALYSES FOR HANDLING MISSING DATA

The investigators aim to collect the baseline characteristics and follow-up parameters on all the participant and control populations in the best possible way. In first instance for prevention of missing data, the missing data will be flagged up in the data entry stage and investigators will try their best to collect this information from the database and patient follow up. The following methods of analyses will be used to handle missing data:

* Complete case analysis: In this analysis the participants with missing data will be excluded from the primary analysis. This will reduce the sample size; however, the observed data will not be biased. The extent of missing data will be reported in the limitations of the study. Complete case analysis will be used as primary analysis in the following situations: Proportion of the missing data are <5% or >40%; certainty that the missing data is completely at random (MCAR) (In MCAR the mechanism causing missing data may depend neither on observed data nor on the missing data); only the dependent variable data is missing and auxiliary variables are not identified
* Multiple imputation: This will be used as primary method to handle the missing data if the above situations are excluded.

CONFIDENTIALITY AND DATA PROTECTION A unique trial identification number will be used for identification of study participants. All the personal data used in the study will be processed in accordance with the Data protection Act 2018 and will be regarded as strictly confidential.

CONFLICTS OF INTEREST There are no conflicts of interest associated with this study.

AMENDMENTS Any amendments to the study protocol or documentation will be initiated by the Chief Investigator. All substantial amendments will be submitted to IRB for approval followed by implementation of the changes in all sites involved in the study. Amendments will be documented in the 'Protocol Amendment' section of the study protocol.

END OF PROJECT DEFINITION Patient recruitment will occur over the course of 18 months. In order to follow up the patients for the outcome of live birth rate, data analysis, manuscript writing, and publication will take place over the subsequent 12 months.

September 2022: Amendments to the protocol: Some of the methodological aspects of the AdAPT-ART study to ensure timely delivery of the study to a full sample size. These amendments have been approved by the ethics committee and are as follows:

1. Removal of patient consent specific to the study and use of HFEA CD form to confirm their consent for participation in research Rationale: A. Data of women undergoing IVF/ICSI who consent for participation in research on the HFEA CD form will be looked at B. Baseline ultrasound scan which is the diagnostic tool for adenomyosis is part of routine management and there is no additional step or intervention involved in the study
2. Eligibility criteria: Amendment added in the eligibility section
3. Sample size: Amendment added in the groups section Rationale: In the preliminary stages we had not realized the uneven balance that exists between patients with normal uterus and those with adenomyosis undergoing ART cycles. Our latest unpublished systematic review on prevalence of adenomyosis in a subgroup of women undergoing ART has concluded the prevalence of 11% which translates to 11 women with adenomyosis to 100 women with normal uterus undergoing ART

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and ≤42 years: Maternal age is an independent factor affecting the live birth rate in ART cycles. In 2019, a steep drop in the live birth rate has been reported in the United Kingdom in the latest Human Fertilisation and Embryology Authority (HFEA) data from the 32% per embryo transferred for patients under 35 years, compared to below 5% for patients aged 43+ when using their own eggs (HFEA, 2021). Hence, this is the age cut-off used in the study.
* Undergoing IVF/ICSI cycle.

Exclusion Criteria:

* Coexisting fibroid uterus. The sensitivity of TVUS for diagnosis of adenomyosis gradually decreases to as low as 33% when fibroids are present (Chapron et al, 2020; Dueholm et al, 2001) and hence this is a reasonable exclusion criterion due to risk of confounding.
* Endometriosis: Endometrioma confirmed on USS or known laparoscopic diagnosis of endometriosis (with histological confirmation). This will not fully exclude endometriosis in all the participants included in the study and inclusion of these potential missed cases of endometriosis will be one of the limiting factors of the study.
* Untreated hydrosalpinx
* Uterine malformation
* Previous myomectomy
* Previous surgery for adenomyosis
* Inconclusive USS

September 2022: Amendments to the protocol: Some of the methodological aspects of the AdAPT-ART study have been revisited to ensure timely delivery of the study to a full sample size and to make the recruitment smooth. These amendments have been approved by the local ethics committee.

Amendment to the eligibility criteria: Inclusion:

1. Age: 18-45 years (Age will be adjusted for)
2. Endometriosis: Subgroup analysis for isolated adenomyosis and those with coexisting endometriosis will be performed

Rationale: Adenomyosis with coexisting endometriosis is common and is an important group to look at in terms of outcome of pregnancy loss.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study cohort will comprise of women diagnosed with adenomyosis on pre-treatment baseline ultrasound scan before ART treatment who satisfy the eligibility criteria and consent to participate in the study. The Morphological Uterus Sonographic Assessment (MUSA) criteria will be used to describe the ultrasound features of adenomyosis. The MUSA criteria outlines the ultrasound features of myometrium and myometrial lesions using standardised terms, definitions and measurements. A diagnosis of adenomyosis is made if any morphological features of adenomyosis are present.
Sampling Method: Non-Probability Sample
Enrollment: 828 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pregnancy loss at <24 weeks gestation | up to 24 weeks gestation
  Pregnancy loss up to 24 weeks out of all pregnancies achieved. The pregnancy loss will include biochemical pregnancy loss, miscarriage, pregnancy of unknown location (PUL) and ectopic pregnancy.1. Biochemical pregnancy: Spontaneous pregnancy demise based on a previous positive pregnancy test that then becomes negative without an ultrasound evaluation 2. Miscarriage: Intrauterine pregnancy demise confirmed by TVS or histology of pregnancy tissue. This would be before 24 completed weeks of gestational age. The gestational age limit is based on the legal viability limit in the United Kingdom.
  3. Pregnancy of unknown location (PUL): Temporary classification to describe when no pregnancy can be visualised inside or outside the uterus on TVS in a woman with a positive pregnancy test.

SECONDARY OUTCOMES:
Number of gestational sacs observed at vaginal ultrasound 3-5 weeks after transfer per embryo transfer | 3-5 weeks after transfer
  Implantation rate per embryo transfer and per woman: Number of gestational sacs divided by number of embryos transferred
Number of participants with positive pregnancy test following embryo transfer | 14-16 days after embryo transfer
  Biochemical pregnancy rate per embryo transfer: Positive pregnancy test following embryo transfer
Number of participants with clinical pregnancy per embryo transfer | 6-7 weeks gestation
  Presence of at least one intrauterine gestational sac on ultrasound
Number of participants with ongoing pregnancy | 12 weeks gestation
  Defined as a live pregnancy at 12 weeks onwards
Number of participants with live birth | 34 weeks gestation
  Live birth rate after 34 weeks per woman

CONTACTS AND LOCATIONS:
Overall Officials: Arri Coomarasamy, Study Director — University of Birmingham
Locations (9):
- United Kingdom (9):
  - CARE Fertility, Birmingham, Birmingham, England
  - CARE Fertility, Chester, Chester, England
  - CARE Fertility, Manchester, Manchester, England
  - CARE Fertility, Nottingham, Nottingham, England
  - CARE Fertility, Sheffield, Sheffield, England
  - CARE Fertility, Tamworth, Tamworth, England
  - CARE Fertility Bolton, Bolton
  - CARE Fertility, Leeds, Leeds
  - CARE Fertility, Northampton, Northampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andres MP, Borrelli GM, Ribeiro J, Baracat EC, Abrao MS, Kho RM. Transvaginal Ultrasound for the Diagnosis of Adenomyosis: Systematic Review and Meta-Analysis. J Minim Invasive Gynecol. 2018 Feb;25(2):257-264. doi: 10.1016/j.jmig.2017.08.653. Epub 2017 Aug 30. PMID 28864044
- [Background] Chapron C, Vannuccini S, Santulli P, Abrao MS, Carmona F, Fraser IS, Gordts S, Guo SW, Just PA, Noel JC, Pistofidis G, Van den Bosch T, Petraglia F. Diagnosing adenomyosis: an integrated clinical and imaging approach. Hum Reprod Update. 2020 Apr 15;26(3):392-411. doi: 10.1093/humupd/dmz049. PMID 32097456
- [Background] Chiang CH, Chang MY, Shiau CS, Hou HC, Hsieh TT, Soong YK. Effect of a sonographically diffusely enlarged uterus without distinct uterine masses on the outcome of in vitro fertilization-embryo transfer. J Assist Reprod Genet. 1999 Aug;16(7):369-72. doi: 10.1023/a:1020593930366. PMID 10459520
- [Background] Dueholm M, Lundorf E, Hansen ES, Sorensen JS, Ledertoug S, Olesen F. Magnetic resonance imaging and transvaginal ultrasonography for the diagnosis of adenomyosis. Fertil Steril. 2001 Sep;76(3):588-94. doi: 10.1016/s0015-0282(01)01962-8. PMID 11532486
- [Background] Exacoustos C, Brienza L, Di Giovanni A, Szabolcs B, Romanini ME, Zupi E, Arduini D. Adenomyosis: three-dimensional sonographic findings of the junctional zone and correlation with histology. Ultrasound Obstet Gynecol. 2011 Apr;37(4):471-9. doi: 10.1002/uog.8900. PMID 21433167
- [Background] Exacoustos C, Morosetti G, Conway F, Camilli S, Martire FG, Lazzeri L, Piccione E, Zupi E. New Sonographic Classification of Adenomyosis: Do Type and Degree of Adenomyosis Correlate to Severity of Symptoms? J Minim Invasive Gynecol. 2020 Sep-Oct;27(6):1308-1315. doi: 10.1016/j.jmig.2019.09.788. Epub 2019 Oct 7. PMID 31600574
- [Background] Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials - a practical guide with flowcharts. BMC Med Res Methodol. 2017 Dec 6;17(1):162. doi: 10.1186/s12874-017-0442-1. PMID 29207961
- [Background] Human Fertilisation and Embryology Authority (HFEA). Fertility-treatment 2019: trends and figures. UK statistics for IVF and DI treatment, storage, and donation. May 2021. Available from: Fertility treatment 2019: trends and figures | Human Fertilisation and Embryology Authority (hfea.gov.uk) [Accessed 12th July 2021]
- [Background] Huang Y, Zhao X, Chen Y, Wang J, Zheng W, Cao L. Miscarriage on Endometriosis and Adenomyosis in Women by Assisted Reproductive Technology or with Spontaneous Conception: A Systematic Review and Meta-Analysis. Biomed Res Int. 2020 Dec 8;2020:4381346. doi: 10.1155/2020/4381346. eCollection 2020. PMID 33490243
- [Background] Lazzeri L, Morosetti G, Centini G, Monti G, Zupi E, Piccione E, Exacoustos C. A sonographic classification of adenomyosis: interobserver reproducibility in the evaluation of type and degree of the myometrial involvement. Fertil Steril. 2018 Nov;110(6):1154-1161.e3. doi: 10.1016/j.fertnstert.2018.06.031. PMID 30396560
- [Background] Maheshwari A, Gurunath S, Fatima F, Bhattacharya S. Adenomyosis and subfertility: a systematic review of prevalence, diagnosis, treatment and fertility outcomes. Hum Reprod Update. 2012 Jul;18(4):374-92. doi: 10.1093/humupd/dms006. Epub 2012 Mar 22. PMID 22442261
- [Background] Munro MG. Uterine polyps, adenomyosis, leiomyomas, and endometrial receptivity. Fertil Steril. 2019 Apr;111(4):629-640. doi: 10.1016/j.fertnstert.2019.02.008. PMID 30929720
- [Background] Naftalin J, Hoo W, Nunes N, Mavrelos D, Nicks H, Jurkovic D. Inter- and intraobserver variability in three-dimensional ultrasound assessment of the endometrial-myometrial junction and factors affecting its visualization. Ultrasound Obstet Gynecol. 2012 May;39(5):587-91. doi: 10.1002/uog.10133. PMID 22045594
- [Background] Neal S, Morin S, Werner M, Gueye NA, Pirtea P, Patounakis G, Scott R Jr, Goodman L. Three-dimensional ultrasound diagnosis of adenomyosis is not associated with adverse pregnancy outcome following single thawed euploid blastocyst transfer: prospective cohort study. Ultrasound Obstet Gynecol. 2020 Oct;56(4):611-617. doi: 10.1002/uog.22065. PMID 32349167
- [Background] Pinzauti S, Lazzeri L, Tosti C, Centini G, Orlandini C, Luisi S, Zupi E, Exacoustos C, Petraglia F. Transvaginal sonographic features of diffuse adenomyosis in 18-30-year-old nulligravid women without endometriosis: association with symptoms. Ultrasound Obstet Gynecol. 2015 Dec;46(6):730-6. doi: 10.1002/uog.14834. PMID 25728241
- [Background] Quenby S, Gallos ID, Dhillon-Smith RK, Podesek M, Stephenson MD, Fisher J, Brosens JJ, Brewin J, Ramhorst R, Lucas ES, McCoy RC, Anderson R, Daher S, Regan L, Al-Memar M, Bourne T, MacIntyre DA, Rai R, Christiansen OB, Sugiura-Ogasawara M, Odendaal J, Devall AJ, Bennett PR, Petrou S, Coomarasamy A. Miscarriage matters: the epidemiological, physical, psychological, and economic costs of early pregnancy loss. Lancet. 2021 May 1;397(10285):1658-1667. doi: 10.1016/S0140-6736(21)00682-6. Epub 2021 Apr 27. PMID 33915094
- [Background] Rasmussen CK, Hansen ES, Dueholm M. Inter-rater agreement in the diagnosis of adenomyosis by 2- and 3-dimensional transvaginal ultrasonography. J Ultrasound Med. 2019 Mar;38(3):657-666. doi: 10.1002/jum.14735. Epub 2018 Sep 4. PMID 30182497
- [Background] ESHRE Guideline Group on RPL; Bender Atik R, Christiansen OB, Elson J, Kolte AM, Lewis S, Middeldorp S, Nelen W, Peramo B, Quenby S, Vermeulen N, Goddijn M. ESHRE guideline: recurrent pregnancy loss. Hum Reprod Open. 2018 Apr 6;2018(2):hoy004. doi: 10.1093/hropen/hoy004. eCollection 2018. PMID 31486805
- [Background] Sun YL, Wang CB, Lee CY, Wun TH, Lin P, Lin YH, Tseng CC, Chen CH, Tseng CJ. Transvaginal sonographic criteria for the diagnosis of adenomyosis based on histopathologic correlation. Taiwan J Obstet Gynecol. 2010 Mar;49(1):40-4. doi: 10.1016/S1028-4559(10)60007-1. PMID 20466291
- [Background] Tummers P, De Sutter P, Dhont M. Risk of spontaneous abortion in singleton and twin pregnancies after IVF/ICSI. Hum Reprod. 2003 Aug;18(8):1720-3. doi: 10.1093/humrep/deg308. PMID 12871890
- [Background] Van den Bosch T, de Bruijn AM, de Leeuw RA, Dueholm M, Exacoustos C, Valentin L, Bourne T, Timmerman D, Huirne JAF. Sonographic classification and reporting system for diagnosing adenomyosis. Ultrasound Obstet Gynecol. 2019 May;53(5):576-582. doi: 10.1002/uog.19096. No abstract available. PMID 29790217
- [Background] Van den Bosch T, Dueholm M, Leone FP, Valentin L, Rasmussen CK, Votino A, Van Schoubroeck D, Landolfo C, Installe AJ, Guerriero S, Exacoustos C, Gordts S, Benacerraf B, D'Hooghe T, De Moor B, Brolmann H, Goldstein S, Epstein E, Bourne T, Timmerman D. Terms, definitions and measurements to describe sonographic features of myometrium and uterine masses: a consensus opinion from the Morphological Uterus Sonographic Assessment (MUSA) group. Ultrasound Obstet Gynecol. 2015 Sep;46(3):284-98. doi: 10.1002/uog.14806. Epub 2015 Aug 10. PMID 25652685
- [Background] Vercellini P, Consonni D, Dridi D, Bracco B, Frattaruolo MP, Somigliana E. Uterine adenomyosis and in vitro fertilization outcome: a systematic review and meta-analysis. Hum Reprod. 2014 May;29(5):964-77. doi: 10.1093/humrep/deu041. Epub 2014 Mar 12. PMID 24622619
- [Background] Younes G, Tulandi T. Effects of adenomyosis on in vitro fertilization treatment outcomes: a meta-analysis. Fertil Steril. 2017 Sep;108(3):483-490.e3. doi: 10.1016/j.fertnstert.2017.06.025. PMID 28865548
- [Background] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Hum Reprod. 2017 Sep 1;32(9):1786-1801. doi: 10.1093/humrep/dex234. PMID 29117321